CLINICAL TRIAL: NCT04875429
Title: Zenith® Fenestrated+ Endovascular Graft Clinical Study
Brief Title: Zenith® Fenestrated+ Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-07
Record Dates: First submitted 2021-04-19; First posted 2021-05-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aortic Aneurysm, Abdominal; Juxtarenal Aortic Aneurysm; Extent IV Thoracoabdominal; Pararenal Aneurysm
Keywords: endovascular; Vascular Diseases; Cardiovascular Diseases; Fenestration
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aortic abdominal aneurysm (Experimental)
  Interventions: Device: Zenith Fenestrated+ Endovascular Graft in combination with the BeGraft Balloon-Expandable FEVAR Bridging Stent Graft System and Unibody2

INTERVENTIONS:
Device: Zenith Fenestrated+ Endovascular Graft in combination with the BeGraft Balloon-Expandable FEVAR Bridging Stent Graft System and Unibody2 — Endovascular aneurysm repair

SUMMARY:
The Zenith® Fenestrated+ Endovascular Graft Clinical Study will assess the safety and effectiveness of the Zenith® Fenestrated+ Endovascular Graft (ZFEN+) in combination with the BeGraft Balloon-Expandable FEVAR Bridging Stent Graft System (BeGraft) and Unibody2 for the treatment of patients with aortic aneurysms involving one or more of the major visceral arteries.

ELIGIBILITY:
Include Criteria:

1. Thoracoabdominal, pararenal or juxtarenal aortic aneurysm with a diameter ≥ 55 mm for males and ≥ 50 mm for females
2. Thoracoabdominal, pararenal or juxtarenal aortic aneurysm with a growth rate of ≥ 5 mm in 6 months
3. Thoracoabdominal, pararenal or juxtarenal aortic aneurysm with aortic diameter > 2x the normal aortic diameter or saccular aneurysm that warrants treatment in the opinion of the investigator

Exclusion Criteria:

1. Age < 18 years
2. Life expectancy < 2 years
3. Pregnant, breast-feeding, or planning to become pregnant within 60 months
4. Inability or refusal to give informed consent by the patient or legally authorized representative
5. Unwilling or unable to comply with the follow-up schedule, required clinical assessments, and imaging
6. Simultaneous participation in another investigation study, unless the patient is at least 30 days beyond the primary endpoint of any previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Composite measure of device technical success and procedural safety | 30 days post procedure
  Percent of patients with device technical success and freedom from procedural safety events in the following criteria:
  1. Device technical success which includes delivery, deployment, and withdrawal of the device without the need for unanticipated corrective intervention), and
  2. Freedom from the following procedural safety events: rupture, aneurysm-related mortality, permanent paraplegia, new onset renal failure requiring dialysis, bowel ischemia requiring surgery, and disabling stroke
Composite measure of freedom from aneurysm-related mortality and clinically significant reintervention | 12 months post procedure
  Percent of patients meeting the following criteria:
  1. Freedom from aneurysm-related mortality (death from aneurysm rupture, death from any cause occurring within 30 days of procedure or secondary intervention or device or procedure related death) and
  2. Freedom from clinically significant reintervention (including open surgery to restore blood flow or restore bodily function, any device related intervention requiring hospitalization, placement of an additional endovascular graft component(s), placement of a stent(s) as indicated for loss of or for having inadequate fixation, seal or patency)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Oderich, MD, Principal Investigator — Baylor College of Medicine
Locations (33):
- United States (32):
  - University of Alabama Birmingham Hospital, Birmingham, Alabama
  - UC San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Shands Hospital, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Endeavor Health Cardiovascular Institute at Glenbrook Hospital, Glenview, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital, Naperville, Illinois
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York University Langone Medical Center, New York, New York
  - Columbia University Irving Medical Center/NY Presbyterian Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Holston Valley Hospital, Kingsport, Tennessee
  - Ut Southwestern, Dallas, Texas
  - Memorial Hermann Texas Medical Center/UT Health, Houston, Texas
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after publication of the results from this study and ending 5 years after initial publication. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.